CLINICAL TRIAL: NCT04414280
Title: The Impact of Hybrid Closed-loop Insulin Delivery (Medtronic MiniMed 670G and 780G System, and Tandem t:Slim X2 Control-IQ) on Glycemic Control and Patient-reported Outcomes in People Living With Type 1 Diabetes: a Multicenter Real-world Observational Study in Belgium
Brief Title: The Impact of Hybrid Closed-loop Insulin Delivery in Type 1 Diabetes on Glycemic Control and PROMs
Acronym: INRANGE
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof dr Pieter Gillard, Clinical Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S63351
Record Dates: First submitted 2020-04-10; First posted 2020-06-04 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Hybrid closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- type 1 diabetes patients using Medtronic MiniMed 670G: Patients with type 1 diabetes, aged 8 years or older, who start with the Medtronic MiniMed 670G system (as part of routine clinical practice) in one of the 17 participating centers and who signed informed consent are eligible to participate. The decision about which patient to start, is left to the clinical judgement of the treating health care professional.
  Interventions: Device: Medtronic MiniMed 670G
- type 1 diabetes patients using Medtronic MiniMed 780G: Patients with type 1 diabetes, aged 8 years or older, who start with the Medtronic MiniMed 780G system (as part of routine clinical practice) in one of the 17 participating centers and who signed informed consent are eligible to participate. The decision about which patient to start, is left to the clinical judgement of the treating health care professional.
  Interventions: Device: Medtronic MiniMed 780G
- type 1 diabetes patients using Tandem Control-IQ: Patients with type 1 diabetes, aged 6 years or older, who start with the Tandem Control-IQ system (as part of routine clinical practice) in one of the 17 participating centers and who signed informed consent are eligible to participate. The decision about which patient to start, is left to the clinical judgement of the treating health care professional.
  Interventions: Device: Tandem Control-IQ

INTERVENTIONS:
Device: Medtronic MiniMed 670G — The Medtronic Minimed 670G system is a form of hybrid closed-loop insulin delivery. The Medtronic MiniMed 670G system automatically adjusts basal insulin every five minutes based on CGM readings to reach a glucose target of 120 mg/dL, the SmartGuard Auto Mode. Patients still need to enter their carbohydrate intake and administer meal-time and correction boluses. Before Auto Mode is introduced, the Medtronic MiniMed 670G system has to be worn in Manual Mode. In contrast to Auto Mode, Manual Mode features an insulin stop up to 30 minutes before or when reaching preset low limits (suspend before/on low) and an automatic insulin restart when blood sugar levels recover. During Manual Mode the pump 'becomes familiar with' the daily insulin need of the patient. This information will be used when in Auto Mode.
  Groups: type 1 diabetes patients using Medtronic MiniMed 670G
Device: Medtronic MiniMed 780G — The Medtronic Minimed 780G system differs in several aspects from the MiniMed 670G system. In Auto Mode, the user can choose from two target levels for even more stricter glucose control (100 mg/dL and 120 mg/dL) and correction boluses are now automated without the need of user interaction. When administering meal boluses, no capillary blood glucose value is required. The safety feature to exit from Auto Mode to Manual Mode was too strict in the Minimed 670G. In the Minimed 780G this is more flexible to overcome this frequently reported patient frustration.
  Groups: type 1 diabetes patients using Medtronic MiniMed 780G
Device: Tandem Control-IQ — The Tandem t:slim X2 Control-IQ consists of the Tandem t:slim X2 insulin pump with Control-IQ technology, and integrates with the Dexcom G6 CGM-device via Bluetooth. Blood glucose readings for calibration are not required. The Tandem t:slim X2 Control-IQ automatically adjusts basal insulin based on CGM readings to reach a glucose target range between of 112-160 mg/dL. Patients still need to enter their carbohydrate intake and administer meal-time boluses, but the system automatically increases the basal insulin dose or gives automated correction boluses in case of high blood glucose levels. The technology offers optional settings for sleep and exercise, with different glucose targets in order to match the insulin need during these activities. New versions of the pump software can be downloaded and installed remotely via the user's own computer.
  Groups: type 1 diabetes patients using Tandem Control-IQ

SUMMARY:
Since February 2019 the first hybrid closed-loop insulin pump, the Medtronic MiniMed 670G system, has been offered to people with type 1 diabetes in Belgium. Despite previous studies, the impact of these new kinds of insulin pumps on glycemic control and patient-reported outcomes (PROMs) is still unclear. Therefore, this study will evaluate the impact of the Medtronic MiniMed 670G, Medtronic MiniMed 780G and Tandem Control-IQ systems on glycemic control and PROMs in people living with type 1 diabetes under real-life conditions. In a multicenter real-world observational study, 350 adults and 100 children with type 1 diabetes who are treated with each of these systems in one of 17 Belgian centers, will be followed for a period of 24 months. The primary endpoint is the evolution of time spent in range (defined as a sensor glucose value between 70 and 180 mg/dL) from before start to 12 months after start of hybrid closed-loop therapy.

Since not much is known about the impact of hybrid closed-loop on partners of adults living with type 1 diabetes, an optional substudy (INRANGE-PARTNER) will be performed investigating the quality of life in partners of adults of type 1 diabetes using hybrid closed-loop therapy. More specifically, the substudy will compare the quality of life of partners of type 1 diabetes patients both before and after implementation of hybrid closed-loop therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 diabetes
* patients aged 6 years or older
* patients starting with hybrid closed-loop therapy (as part of routine clinical practice) in one of the 17 participating centers. Note: the decision about which patient to start, is left to the clinical judgement of the treating health care professional.
* patients who signed informed consent

Exclusion Criteria:

* patients without type 1 diabetes
* patients under 6 years of age
* patients not starting with hybrid closed-loop therapy in one of the 17 participating centers
* patients who did not sign informed consent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited at the Diabetes departments of 17 diabetes convention hospitals in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in range | 12 months
  The evolution of percentage of time spent in range (sensor glucose 70-180 mg/dL) from before start to 12 months after start

SECONDARY OUTCOMES:
Time in range | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent in range (sensor glucose 70-180 mg/dL), with exclusion of the primary endpoint
Time in level 2 hypoglycemia | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent in level 2 hypoglycemia (sensor glucose <54 mg/dL)
Time in level 1 hypoglycemia | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent in level 1 hypoglycemia (sensor glucose <70 mg/dL and ≥54 mg/dL)
Time below range | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent below range (sensor glucose <70 mg/dL)
Time above range | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent above range (sensor glucose >180 mg/dL)
Time in level 1 hyperglycemia | from before start to 4, 8, 12 and 24 months after start
  Percentage of time spent in level 1 hyperglycemia (sensor glucose >250 mg/dL)
Glycemic variability | from before start to 4, 8, 12 and 24 months after start
  Glycemic variability: coefficient of variation (CV), standard deviation (SD) and mean amplitude of glycemic excursions (MAGE)
Mean glucose concentration | from before start to 4, 8, 12 and 24 months after start
  Mean glucose concentration
HbA1c | from before start to 4, 8, 12 and 24 months after start
  Change in HbA1c
Correlation between sex (male/female) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between sex (male/female) and change in HbA1c
Correlation between educational attainment (measured by a questionnaire with multiple options) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between educational attainment (measured by a questionnaire with multiple options) and change in HbA1c
Correlation between cohabitation (yes/no) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between cohabitation (yes/no) and change in HbA1c
Correlation between duration of diabetes (years) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between duration of diabetes (years) and change in HbA1c
Correlation between chronic diabetic complications (measured by a questionnaire with multiple options) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between chronic diabetic complications (measured by a questionnaire with multiple options) and change in HbA1c
Correlation between total daily dose of insulin (units per day) and change in HbA1c | from before start to 4, 8, 12 and 24 months after start
  Correlation between total daily dose of insulin (units per day) and change in HbA1c
Number of low glucose events | from before start to 4, 8, 12 and 24 months after start
  Number of low glucose events (LGE, defined as sensor glucose values ≤54 mg/dL for at least 15 minutes, preceded by at least 30 minutes with sensor glucose values >54 mg/dL)
Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire (scale: 0 (low quality of life) - 100 (high quality of life)) | from before start to 4, 8, 12 and 24 months after start for adults
  Quality of life measured by the Short Form Health Survey 36-item (SF-36) version 2 questionnaire (scale: 0 (low quality of life) - 100 (high quality of life))
Hypoglycemia awareness measured by the Clarke hypoglycemia awareness survey (scale: unaware (≥4 times "R" or once "U") or aware (<4 times "R")) | from before start to 4, 8, 12 and 24 months after start for adults and children
  Hypoglycemia awareness measured by the Clarke hypoglycemia awareness survey (scale: unaware (≥4 times "R" or once "U") or aware (<4 times "R"))
Hypoglycemia awareness measured by the Gold-scale (scale: 1 (aware) - 7 (unaware)) | from before start to 4, 8, 12 and 24 months after start for adults and children
  Hypoglycemia awareness measured by the Gold-scale (scale: 1 (aware) - 7 (unaware))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, behaviour (scale: 0 (less adapted behaviour) - 40 (more adapted behaviour)) | from before start to 4, 8, 12 and 24 months after start for adults
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, behaviour (scale: 0 (less adapted behaviour) - 40 (more adapted behaviour))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry (scale: 0 (not worried) - 72 (very worried)) | from before start to 4, 8, 12 and 24 months after start for adults
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey, version II (HFS-II) questionnaire, worry (scale: 0 (not worried) - 72 (very worried))
Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire (scale: 0 (no distress) - 20 (very distressed)) | from before start to 4, 8, 12 and 24 months after start for adults
  Distress due to diabetes measured by the Problem Areas In Diabetes survey, short form (PAID-SF) questionnaire (scale: 0 (no distress) - 20 (very distressed))
Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire, status (DTSQs. Scale: 0 (low satisfaction) - 36 (high satisfaction)) | from before start to 4, 8, 12 and 24 months after start for adults
  Treatment satisfaction measured by the Diabetes Treatment Satisfaction Questionnaire, status (DTSQs. Scale: 0 (low satisfaction) - 36 (high satisfaction))
Treatment satisfaction measured by a self-developed questionnaire about expectations towards the use of the Medtronic MiniMed 670G system (multiple choice) | at 4, 8, 12 and 24 months after start of the Medtronic MiniMed 670G and 780G system for adults and children
  Treatment satisfaction measured by a self-developed questionnaire about expectations towards the use of the Medtronic MiniMed 670G system (multiple choice)
Impact of diabetes and device satisfaction by the Diabetes Impact and Device Satisfaction Scale (scale: device satisfaction = 7 (not satisfied) - 70 (very satisfied); diabetes impact = 4 (low impact) - 40 (high impact)) | from before start to 4, 8, 12 and 24 months after start of the Tandem Control-IQ for adults
  Impact of diabetes and device satisfaction by the Diabetes Impact and Device Satisfaction Scale (scale: device satisfaction = 7 (not satisfied) - 70 (very satisfied); diabetes impact = 4 (low impact) - 40 (high impact))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey for children (HFS-C) questionnaire, worry (scale: 0 (not worried) - 60 (very worried)) | from before start to 4, 8, 12 and 24 months after start of the Tandem Control-IQ for children
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey for children (HFS-C) questionnaire, worry (scale: 0 (not worried) - 60 (very worried))
Fear of hypoglycemia measured by the Hypoglycemia Fear Survey for children (HFS-C) questionnaire, behaviour (scale: 0 (less adapted behaviour) - 40 (more adapted behaviour)) | from before start to 4, 8, 12 and 24 months after start for children
  Fear of hypoglycemia measured by the Hypoglycemia Fear Survey for children (HFS-C) questionnaire, behaviour (scale: 0 (less adapted behaviour) - 40 (more adapted behaviour))
The Diabetes Quality of Life for Youth (DQOLY) questionnaire | from before start to 4, 8, 12 and 24 months after start for children
  The Diabetes Quality of Life for Youth (DQOLY) questionnaire
Questionnaire for parents of children and adolescents with diabetes, a part of the HAPPI-D QOL Protocol (Hvidøre, Adolescent, Parent, Professional, Instrument, Diabetes) | from before start to 4, 8, 12 and 24 months after start for parents
  Questionnaire for parents of children and adolescents with diabetes, a part of the HAPPI-D QOL Protocol (Hvidøre, Adolescent, Parent, Professional, Instrument, Diabetes)
The Parent's fear of hypoglycemia scale - modified version of the Hypoglycemia Fear Survey for use with parents | from before start to 4, 8, 12 and 24 months after start for parents
  The Parent's fear of hypoglycemia scale - modified version of the Hypoglycemia Fear Survey for use with parents

OTHER OUTCOMES:
Composite endpoint of HbA1c and time in hypoglycemia <70 mg/dl | from before start to 4, 8, 12 and 24 months after start
  Composite endpoint of HbA1c and time in hypoglycemia <70 mg/dl
Severe hypoglycemia | from before start to 4, 8, 12 and 24 months after start
  Frequency of severe hypoglycemia
Diabetic ketoacidosis | from before start to 4, 8, 12 and 24 months after start
  Frequency of diabetic ketoacidosis
Hospital visits and/or admissions | from before start to 4, 8, 12 and 24 months after start
  Number of hospital visits and/or admissions because of severe hypoglycemia or diabetic ketoacidosis
Work and school absenteeism | from before start to 4, 8, 12 and 24 months after start
  Work and school absenteeism (number of days that a patient was unable to attend work/school due to his/her diabetes (excluding consultation))
(Unplanned) contacts with the diabetes team | from before start to 4, 8, 12 and 24 months after start
  Frequency of (unplanned) contacts with the diabetes team
Change in total daily dose of insulin (units/day) | from before start to 4, 8, 12 and 24 months after start
  Change in total daily dose of insulin (units/day)
Change in body weight (kilograms) | from before start to 4, 8, 12 and 24 months after start
  Change in body weight (kilograms)
Time in Manual Mode | only measured at month 4, 8, 12 and 24 after start of the Medtronic MiniMed 670G an 780G system
  Percentage of time spent in Manual Mode
Time in Auto Mode | only measured at month 4, 8, 12 and 24 after start of the Medtronic MiniMed 670G an 780G system
  Percentage of time spent in Auto Mode
Indications for use of hybrid closed-loop therapy measured by a self-developed questionnaire (multiple options (non-ordinal)) | at start
  Indications for use of hybrid closed-loop therapy measured by a self-developed questionnaire (multiple options (non-ordinal))
Patients who stop | only measured at stop
  Number of patients who stop with hybrid closed-loop therapy
Reasons for discontinuation of hybrid closed-loop therapy measured by a self-developed questionnaire (multiple choice) | only measured at stop
  Reasons for discontinuation of hybrid closed-loop therapy measured by a self-developed questionnaire (multiple choice)
Quality of life in partners of T1D patients using hybrid closed-loop therapy measured by the SF-36 version 2 questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Quality of life in partners of T1D patients using hybrid closed-loop therapy measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Quality of life in partners of T1D patients using hybrid closed-loop therapy measured by the DIDP-FM questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Quality of life in partners of T1D patients using hybrid closed-loop therapy measured by the DAWN (Diabetes Attitudes, Wishes and Needs) Impact of Diabetes Profile Family Members (DIDP-FM) questionnaire (scale: 0 (less negative impact) - 100 (more negative impact)) Note: only in case of substudy
Difference in quality of life in partners of T1D patients before and after implementation of hybrid closed-loop therapy, measured by the SF-36 version 2 questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Difference in quality of life in partners of T1D patients before and after implementation of hybrid closed-loop therapy, measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Difference in quality of life in partners of T1D patients before and after implementation of hybrid closed-loop therapy, measured by the DIDP-FM questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Difference in quality of life in partners of T1D patients before and after implementation of hybrid closed-loop therapy, measured by the DIDP-FM questionnaire. Note: only in case of substudy
Correlation between 'quality of life of T1D patients using hybrid closed-loop therapy' and 'quality of life in partners of T1D patients', both measured by the SF-36 version 2 questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'quality of life of T1D patients using hybrid closed-loop therapy' and 'quality of life in partners of T1D patients', both measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Correlation between composite endpoint 'HbA1c and time in hypoglycemia <70 mg/dL' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2. Note: substudy only | from before start to 12 months after start
  Correlation between composite endpoint 'HbA1c and time in hypoglycemia <70 mg/dL' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Correlation between composite endpoint 'HbA1c and time in hypoglycemia <70 mg/dL' and 'quality of life in partners of T1D patients using the hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: substudy only | from before start to 12 months after start
  Correlation between composite endpoint 'HbA1c and time in hypoglycemia <70 mg/dL' and 'quality of life in partners of T1D patients using the hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy
Correlation between 'frequency of severe hypoglycemia' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'frequency of severe hypoglycemia' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Correlation between 'frequency of severe hypoglycemia' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'frequency of severe hypoglycemia' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy
Correlation between 'frequency of diabetic ketoacidosis' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'frequency of diabetic ketoacidosis' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Correlation between 'frequency of diabetic ketoacidosis' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'frequency of diabetic ketoacidosis' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy
Correlation between 'duration of type 1 diabetes of the patient (years)' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2. Note: substudy only | from before start to 12 months after start
  Correlation between 'duration of type 1 diabetes of the patient (years)' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the SF-36 version 2 questionnaire. Note: only in case of substudy
Correlation between 'duration of type 1 diabetes of the patient (years)' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy | from before start to 12 months after start
  Correlation between 'duration of type 1 diabetes of the patient (years)' and 'quality of life in partners of T1D patients using hybrid closed-loop therapy', the latter being measured by the DIDP-FM questionnaire. Note: only in case of substudy

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Gillard, MD, Principal Investigator — UZ Leuven
Locations (18):
- Belgium (18):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - OLVZ Aalst, Aalst
  - GZA Ziekenhuizen - campus Sint-Vincentius, Antwerp
  - Hôpital d'Arlon, Arlon
  - Imeldaziekenhuis, Bonheiden
  - AZ Sint-Jan - campus Sint-Jan, Bruges
  - Hôpital Erasme, Brussels
  - UZ Antwerpen, Edegem
  - ZOL - campus Sint-Jan, Genk
  - Jessa Ziekenhuis - campus Salvator, Hasselt
  - UZ Brussel, Jette
  - AZ Groeninge - campus kennedylaan, Kortrijk
  - CHR de La Citadelle, Liège
  - CHU de Liège - site du Sart Tilman, Liège
  - Az Damiaan, Ostend
  - AZ Delta - campus Wilgenstraat Roeselare, Roeselare
  - AZ Nikolaas, Sint-Niklaas
  - GZA Ziekenhuizen - campus Sint-Augustinus, Wilrijk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Meulemeester J, Keymeulen B, De Block C, Van Huffel L, Taes Y, Ballaux D, Spincemaille K, Lapauw B, Vanhaverbeke G, Lowyck I, Vercammen C, Colin IM, Preumont V, Charleer S, Fieuws S, Mathieu C, Gillard P. One-year real-world benefits of Tandem Control-IQ technology on glucose management and person-reported outcomes in adults with type 1 diabetes: a prospective observational cohort study. Diabetologia. 2025 May;68(5):948-960. doi: 10.1007/s00125-025-06366-x. Epub 2025 Feb 11. PMID 39934368